CLINICAL TRIAL: NCT06612411
Title: Purine Starvation Driven by Host-microbiota Maladaptation Contributes to the Pathogenesis of Irritable Bowel Syndrome
Brief Title: B.Subtilis Attenuate Symptoms in Diarrhea-predominant Irritable Bowel Syndrome by Increasing Hypoxanthine Biosynthesis
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Fangyu Wang, Professor, Jinling Hospital, China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: No.2023DZKY-023-01
Record Dates: First submitted 2024-08-12; First posted 2024-09-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Irritable Bowel Syndrome with Diarrhea; Purine Metabolism Disorder

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- B. subtilis intervention (Active Comparator)
  Interventions: Drug: B. subtilis
- Placebo capsules (Placebo Comparator)
  Interventions: Drug: Dead B. subtilis

INTERVENTIONS:
Drug: B. subtilis — 2 capsules, 3 times a day, orally taken for one month
  Other Names: Medilac-s, S20030087, Beijing Hanmi Pharm.co.,Ltd
  Arms: B. subtilis intervention
Drug: Dead B. subtilis — 2 capsules, 3 times a day, orally taken for one month
  Other Names: Medilac-s, S20030087, Beijing Hanmi Pharm.co.,Ltd
  Arms: Placebo capsules

SUMMARY:
This is a prospective, single-blind, randomized parallel study to investigate whether B. subtilis could improve clinical symptoms of IBS-D patients. Patients are randomly assigned by envelope method. A senior gastroenterologist is responsible for prescribing medication. Researchers are blind to patients' medication. Participants with IBS are recruited and randomized to receive a 4-week administration of B. subtilis-based probiotics. Clinical symptoms and stool samples are collected before and after the trial.

ELIGIBILITY:
Inclusion Criteria:

Patients are diagnosed with IBS. IBS was diagnosed based on the Rome IV criteria. Subjects aged from 16-80 years old without any gut medical conditions like inflammatory bowel diseases, infectious diarrhea, colon tumors were included.

Exclusion Criteria:

Subjects who are taking any probiotics, PPIs, antibiotics or any drugs affecting uric acid levels for at least one month before the study.

Subjects who decline to participate into the study.

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The score of IBS-SSS before and after intervention | 6 months

SECONDARY OUTCOMES:
The concentration of purine in the stool before and after intervention | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Jinling Hospital, Nanjing, China

IPD SHARING:
Plan to Share IPD: Yes